CLINICAL TRIAL: NCT06545032
Title: Minimal Invasive Transforaminal Lumbar Interbody Fusion for Degenerative Lumbar and Lumbosacral Spine Diseases : Clinical and Surgical Outcome
Brief Title: Minimal Invasive Transforaminal Lumbar Interbody Fusion for Degenerative Lumbar and Lumbosacral Spine Diseases
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Abdelaleem Mohamed Abdelrahman, assistant lecturer, Sohag University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: soh-med-24-07-3MD
Record Dates: First submitted 2024-08-06; First posted 2024-08-09 (Actual); Last update posted 2024-08-09 (Actual); Status verified 2024-08

CONDITIONS: Degenerative Spine Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: lumbar fusion — Minimal Invasive Transforaminal Lumbar Interbody Fusion

SUMMARY:
The aim of this study is to evaluate clinical and surgical outcome of MI-TLIF for degenerative lumbar and lumbosacral spine diseases.

DETAILED DESCRIPTION:
Approximately 70% to 85% of adults were affected by low back pain (LBP) at some point during their lifetimes. Numerous anatomic sites can be responsible for the pain, and accurate diagnosis is often difficult. Degenerative lumbar, lumbosacral spine diseases internal disc disruption, lumbar disc herniation, and facet joint arthritis, as well as intra-abdominal pathology, are all potential causes of LBP(Stott and Driscoll, 2024). q Degenerative lumbar and lumbosacral spine diseases are the most rampantly prevalent healthcare problems in the world, with chronic LBP being the second leading cause of adult disability ,The symptoms can broadly be divided into LBP and radicular symptoms in the lower extremities leading in some cases to neurogenic claudication(Shokri et al., 2023).

As an alternative to PLIF, Harms and Rolinger introduced the transforaminal lumbar interbody fusion (TLIF) procedure in 1982 for the management of degenerative spinal disorders that necessitate interbody fusions. The impetus for the development of TLIF was to provide a more lateral approach to the disc space, thus reducing the amount of thecal sac and nerve root retraction. Additionally, in revision cases where scar tissue hinders identification of neural structures, avoidance of midline scar planes with the TLIF procedure is beneficial. Moreover, a circumferential fusion can be achieved from a unilateral approach with the TLIF procedure without having to expose the bilateral epidural space (Karikari, Isaac O. MD; Isaacs, Robert E. MD, 2010).

Technological advances, better magnification and illumination, modern tubular retractors and percutaneous screw systems and more frequent exposure of surgeons to minimally access surgery in their residency training has greatly contributed to the global success of minimal invasive transforaminal lumbar interbody fusion (MI-TLIF). Traditional open spinal fusion surgeries, while effective, are associated with considerable tissue disruption, prolonged recovery times, and higher risks of complications(Prabhu et al., 2022).

MI-TLIFis one such advanced surgical technique designed to treat degenerative conditions of lumbar and lumbosacral spine diseases. Through the tubular expander, MIS-TLIF can reach the facet joints of the diseased segments. MIS-TLIF effectively reduces the peeling and traction injury of the multifidus muscle, prevents postoperative muscle atrophy, and reduces the occurrence of postoperative chronic LBP(Saela et al., 2023).

The MI-TLIF has shown reduced complications, decreased intraoperative blood loss, shorter hospital stays and recovery time, and decreased postoperative narcotic usage while maintaining similar clinical outcomes and fusion rates to conventional open TLIF since its inception (Hong et al., 2022).

The success of MI-TLIF can be attributed to the following fundamental principles: (1) minimizing damage to soft tissues and avoiding destabilization of the spinal segment(s) to achieve the surgical goal with the smallest possible operative footprint; (2) utilizing a unilateral approach to achieve bilateral decompression when needed; and (3) achieving neural decompression indirectly. Although there is no definitive definition of MI-TLIF, the lack of a precise definition has led to significant variations in how surgeons perform the procedure due to various technical nuances associated with each step(Lener et al., 2020).

The use of minimally invasive surgical techniques represents the most recent modification of methods used to achieve lumbar interbody fusion, based upon the premise that a smaller, less traumatic incision should afford better recovery and outcomes(Jang et al., 2024).Hence, in our study we aim to evaluate MI-TLIF for degenerative lumbar and lumbosacral spine diseases.

ELIGIBILITY:
Inclusion Criteria:

* Degenerative spondylolisthesis.
* Degenerative unilateral disc herniations.
* Recurrent disc herniation.

Exclusion Criteria:

* Spondylolisthesis Grade III or IV.
* Degenerative scoliosis .
* Traumatic fracture spine.
* Infections.
* Neoplasms.
* Debilitated patients .
* Coagulation dysfunction.
* Severe osteoporosis.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-09 (Estimated); Primary Completion 2025-09 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
severity of pain according to visual analog score(vas) | 1 year
  comparison between pre & post operative pain

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Fairbank JC, Pynsent PB. The Oswestry Disability Index. Spine (Phila Pa 1976). 2000 Nov 15;25(22):2940-52; discussion 2952. doi: 10.1097/00007632-200011150-00017. PMID 11074683
- [Background] Hong JY, Kim WS, Park J, Kim CH, Jang HD. Comparison of minimally invasive and open TLIF outcomes with more than seven years of follow-up. N Am Spine Soc J. 2022 Jun 11;11:100131. doi: 10.1016/j.xnsj.2022.100131. eCollection 2022 Sep. PMID 35783004
- [Background] Jang HD, Lee JC, Choi SW, Hong CH, Suh YS, Shin BJ. A novel surgical approach using the "lateral corridor" for minimally invasive oblique lumbar interbody fusion at L5-S1: a clinical series and technical note. Eur Spine J. 2024 Jul;33(7):2611-2620. doi: 10.1007/s00586-024-08217-6. Epub 2024 May 31. PMID 38819738
- [Background] Le H, Anderson R, Phan E, Wick J, Barber J, Roberto R, Klineberg E, Javidan Y. Clinical and Radiographic Comparison Between Open Versus Minimally Invasive Transforaminal Lumbar Interbody Fusion With Bilateral Facetectomies. Global Spine J. 2021 Jul;11(6):903-910. doi: 10.1177/2192568220932879. Epub 2020 Jun 22. PMID 32677520